CLINICAL TRIAL: NCT01563991
Title: Impact of Perioperative Intravenous Fluid Utilization on Postoperative Outcomes Following Elective Open Colorectal Surgery
Brief Title: Impact of Perioperative Intravenous Fluid Utilization on Postoperative Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Luca Stocchi, MD, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 07-016
Record Dates: First submitted 2012-03-24; First posted 2012-03-27 (Estimated); Last update posted 2017-03-30 (Actual); Status verified 2017-03

CONDITIONS: Benign Neoplasm of Intestinal Tract; Primary Malignant Neoplasm of Intestinal Tract; Secondary Malignant Neoplasm of Intestinal Tract
Keywords: surgery; fluid; morbidity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard fluid volume (Active Comparator): Subject receives normal fluid volume during peri-operative period
  Interventions: Procedure: Normal fluid volume
- Reduced Fluid Volume (Experimental): Subject receives a reduced fluid volume during the peri-operative period
  Interventions: Procedure: Reduced fluid volume

INTERVENTIONS:
Procedure: Normal fluid volume — Normal fluid group will receive lactated ringes at 8 cc / Kg/ hr total
  Arms: Standard fluid volume
Procedure: Reduced fluid volume — Subject receives 80 cc/ hr LR during the peri-operative period
  Arms: Reduced Fluid Volume

SUMMARY:
Subjects undergoing surgery on the small or large bowel will be randomized to one of 2 groups, a normal fluid amount group and a reduced fluid amount group to evaluate the impact of this change on recovery after surgery.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the impact of reduction in the amount of perioperative fluids on postoperative morbidity, postoperative recovery and the duration of hospitalization. The study will accrue patients undergoing elective open intestinal resection for benign and malignant conditions of the small and large bowel. Patients, who consent to the study, will be randomized at the time of consent, preoperatively. The primary study endpoint will a composite of mortality and major morbidity within the first 30 postoperative days. Secondary endpoints will be return to bowel function (flatus or bowel movement), postoperative hospital stay including the day of surgery and a composite of minor complications. Approximately 186 patients will participate in the study, 93 in each group. Patients will be randomized into one of two groups: the Restricted Fluid Regimen group and the Normal Fluid Administration Regimen group. A very specific flow chart for each group will be followed to distinguish the group. A research nurse will collect the data needed for the study on a daily basis. The patient will be managed by the primary surgeon and his team and the study group flow chart will be followed. If for medical reasons, the patient's care needs to be varied from the study, this is allowed, and will be documented for the study purposes.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years or older
* ASA I-III
* Ability to provide informed consent
* Creatinine less than or equal to 1.3 mg/mL)

Exclusion Criteria:

Patients younger than 18 years old

* ASA IV or higher
* Urgent or emergent surgery
* Mental disease or addictive disorders impairing ability to provide informed consent
* Renal insufficiency (Cr greater than 1.3 mg/mL)
* Significant language barriers
* Cirrhosis causing ascites
* NYHA III or IV, EF less than 25%
* Use of intraoperative epidural anesthesia
* Uncontrolled diabetes
* Uncontrolled hypertension in the opinion of the enrolling surgeon
* ETOH consumption greater than 35 drinks weekly
* Cachexia or absolute neutrophil count of less than 1,200/mm3
* Existing uncontrolled coagulopathy or platelet count of less than 100,000/mm3

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Actual)
Dates: Start 2007-02; Primary Completion 2012-04-18 (Actual); Study Completion 2012-04-18 (Actual)

PRIMARY OUTCOMES:
Morbidity | 5-7 days
  Reduction in post-operative complications at the time of hospital discharge after the surgical episode

CONTACTS AND LOCATIONS:
Overall Officials: Lucci Stocchi, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No